CLINICAL TRIAL: NCT01529749
Title: Effects of Losartan and Antiretroviral Regimen Containing Raltegravir in Fibrosis Inflammation
Brief Title: Effects of Losartan and Antiretroviral Regimen Containing Raltegravir in Fibrosis Inflammation Mediators, Cardiovascular Risk and Neurocognitive Disorders in HIV Infected Patients Previously Effectively Treated
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Felipe Garcia (Other)
Responsible Party: Sponsor-Investigator, Felipe Garcia, Dr, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIV-IMMUNESARTAN; 2011-002071-42 (EudraCT Number)
Record Dates: First submitted 2012-02-08; First posted 2012-02-09 (Estimated); Results first posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-06

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Losartan; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- EFV/FTC/TDF (Active Comparator)
  Interventions: Drug: EFV/FTC/TDF
- EFV/FTC/TDF + Losartan (Experimental)
  Interventions: Drug: EFV/FTC/TDF + Losartan
- FTC/TDF + MK-0518 (Experimental)
  Interventions: Drug: FTC/TDF + MK-0518
- FTC/TDF+MK-0518+Losartan (Experimental)
  Interventions: Drug: FTC/TDF+MK-0518+Losartan

INTERVENTIONS:
Drug: EFV/FTC/TDF + Losartan — EFV/FTC/TDF --> oral, 600/200/245 mg, od Losartan --> initial dose 50 mg/24h, in patients with good tolerance, dose will be increased to 100 mg/24H in week 12.
  Arms: EFV/FTC/TDF + Losartan
Drug: EFV/FTC/TDF — 600/200/245 mg, od, oral
  Arms: EFV/FTC/TDF
Drug: FTC/TDF + MK-0518 — FTC/TDF --> 200/245 mg, oral MK-0518 --> 400 mg, oral
  Arms: FTC/TDF + MK-0518
Drug: FTC/TDF+MK-0518+Losartan — FTC/TDF --> 200/245 mg, oral MK-0518 --> 400 mg, oral Losartan --> -> initial dose 50 mg/24h, in patients with good tolerance, dose will be increased to 100 mg/24n in week 12.
  Arms: FTC/TDF+MK-0518+Losartan

SUMMARY:
This is a open controlled trial in which 48 HIV-1 patients successfully treated with EFV/FTC/TDF will be randomized to one of 4 groups in equal proportion between arms (1:1). The four arms are as follows:

Arm I: EFV / FTC / TDF (n = 12) Arm II: EFV / FTC / TDF + LST (n = 12) Arm III: FTC / TDF + MK-0518 (n = 12) Arm IV: FTC / TDF + LST + MK-0518 (n = 12)

The allocation will take place in two phases:

Phase I: 24 patients 1:1 receiving EFV/FTC/TDF vs. EFV/FTC/TDF + Losartan

If losartan arm shows benefits we will proceed to the second phase:

Phase II: 24 patients 1:1 to receive FTC/TDF+ MK-0518 versus FTC/TDF + MK-0518 + losartan.

Patients will be followed up during 12 months to determinate the proportion of patients with decreased collagen deposition in TL equal to or greater than 50%.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years.
2. Patients with HIV infection in antiretroviral treatment with EFV / FTC / TDF with undetectable viral load (VL <37 copies) for at least 48 weeks.
3. Nadir CD4 +> 250 cells/mm3.
4. Patients, properly informed, give their written consent to participate in the study.

Exclusion Criteria:

1. Criteria for patients with AIDS.
2. Patients with active opportunistic diseases.
3. Patients coinfected with HCV.
4. Patients without tonsillar tissue.
5. Treatment with other drugs receptor antagonists or angiotensin II converting enzyme inhibitors, angiotensin II.
6. Kidney failure.(Glomerular Filtration Rate (GFR < 60 mL/mn)
7. Severe liver failure (PT> 60% ).
8. Pregnant women
9. Known hypersensitivity or contraindication to any study drug.
10. determination of blood pressure (BP) <100/60 mmHg
11. Hyponatremia with serum Na numbers <132 Meq / l
12. History of chronic vomiting the last 6 months
13. History of chronic diarrhea the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-02; Primary Completion 2012-03 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EFV/FTC/TDF | EFV/FTC/TDF + Losartan | FTC/TDF + MK-0518 | FTC/TDF+MK-0518+Losartan
Started | 12 | 12 | 12 | 12
Completed | 12 | 10 | 10 | 10
Not Completed | 0 | 2 | 2 | 2
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EFV/FTC/TDF | EFV/FTC/TDF + Losartan | FTC/TDF + MK-0518 | FTC/TDF+MK-0518+Losartan | Total
Number analyzed (Participants) | 12 | 10 | 10 | 10 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 10 | 10 | 10 | 42
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 40 [33 to 48] | 43 [35 to 49] | 43 [42 to 51] | 35 [32 to 48] | 41 [33 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 0 | 3
  Male | 11 | 8 | 10 | 10 | 39
Region of Enrollment [Number; unit: participants]
  Spain | 12 | 10 | 10 | 10 | 42

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With 50% Reduction of Fibrosis in Lymphatic Tissue.
Time Frame: 48 weeks
Population: Eligibility criteria were being older than 18 years, being on ART with a combined triple therapy regimen and having viral load under the limit of detection for at least the previous 48 weeks.
Measure: Number; unit: participants
Arm/Group | EFV/FTC/TDF | EFV/FTC/TDF + Losartan | FTC/TDF + MK-0518 | FTC/TDF+MK-0518+Losartan
Number analyzed (Participants) | 12 | 10 | 10 | 10
participants | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: EFV/FTC/TDF vs EFV/FTC/TDF + Losartan vs FTC/TDF + MK-0518 vs FTC/TDF+MK-0518+Losartan; Test type: Superiority; p = 1, Chi-squared, Corrected

2. Secondary Outcome: Proportion of Patients With Changes in the Levels of IL-6 in Different Groups.
Time Frame: 48 weeks
Measure: Number; unit: participants
Arm/Group | EFV/FTC/TDF | EFV/FTC/TDF + Losartan | FTC/TDF + MK-0518 | FTC/TDF+MK-0518+Losartan
Number analyzed (Participants) | 12 | 10 | 10 | 10
participants | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: EFV/FTC/TDF vs EFV/FTC/TDF + Losartan vs FTC/TDF + MK-0518 vs FTC/TDF+MK-0518+Losartan; Test type: Superiority; p = 1, Chi-squared, Corrected

3. Secondary Outcome: Proportion of Patients With Changes in the Levels of CRP in Different Groups.
Time Frame: 48 weeks
Measure: Number; unit: participants
Arm/Group | EFV/FTC/TDF | EFV/FTC/TDF + Losartan | FTC/TDF + MK-0518 | FTC/TDF+MK-0518+Losartan
Number analyzed (Participants) | 12 | 10 | 10 | 10
participants | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: EFV/FTC/TDF vs EFV/FTC/TDF + Losartan vs FTC/TDF + MK-0518 vs FTC/TDF+MK-0518+Losartan; Test type: Superiority; p = 1, Chi-squared, Corrected

4. Secondary Outcome: Proportion of Patients With Changes in the Levels of D-dimer in Different Groups.
Time Frame: 48 weeks
Measure: Number; unit: participants
Arm/Group | EFV/FTC/TDF | EFV/FTC/TDF + Losartan | FTC/TDF + MK-0518 | FTC/TDF+MK-0518+Losartan
Number analyzed (Participants) | 12 | 10 | 10 | 10
participants | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: EFV/FTC/TDF vs EFV/FTC/TDF + Losartan vs FTC/TDF + MK-0518 vs FTC/TDF+MK-0518+Losartan; Test type: Superiority; p = 1, Chi-squared, Corrected

5. Secondary Outcome: Proportion of Patients With Increased CD4 in Peripheral Blood.
Time Frame: 48 weeks
Measure: Number; unit: participants
Arm/Group | EFV/FTC/TDF | EFV/FTC/TDF + Losartan | FTC/TDF + MK-0518 | FTC/TDF+MK-0518+Losartan
Number analyzed (Participants) | 12 | 10 | 10 | 10
participants | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: EFV/FTC/TDF vs EFV/FTC/TDF + Losartan vs FTC/TDF + MK-0518 vs FTC/TDF+MK-0518+Losartan; Test type: Superiority; p = 1, Chi-squared, Corrected

6. Secondary Outcome: Proportion of Patients With Increased CD4 in Lymphatic Tissue.
Time Frame: week 48
Measure: Number; unit: participants
Arm/Group | EFV/FTC/TDF | EFV/FTC/TDF + Losartan | FTC/TDF + MK-0518 | FTC/TDF+MK-0518+Losartan
Number analyzed (Participants) | 12 | 10 | 10 | 10
participants | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: EFV/FTC/TDF vs EFV/FTC/TDF + Losartan vs FTC/TDF + MK-0518 vs FTC/TDF+MK-0518+Losartan; Test type: Superiority; p = 1, Chi-squared, Corrected

7. Secondary Outcome: Proportion of Patients With Undetectable Plasma Viral Load in Different Groups
Time Frame: 48 weeks
Measure: Number; unit: participants
Arm/Group | EFV/FTC/TDF | EFV/FTC/TDF + Losartan | FTC/TDF + MK-0518 | FTC/TDF+MK-0518+Losartan
Number analyzed (Participants) | 12 | 10 | 10 | 10
participants | 12 | 10 | 10 | 10
Statistical Analysis 1: Comparison: EFV/FTC/TDF vs EFV/FTC/TDF + Losartan vs FTC/TDF + MK-0518 vs FTC/TDF+MK-0518+Losartan; Test type: Superiority; p = 1, Chi-squared, Corrected

8. Secondary Outcome: Proportion of Patients With Undetectable Viral Load in Lymphatic Tissue in Different Groups
Time Frame: week 48
Measure: Number; unit: participants
Arm/Group | EFV/FTC/TDF | EFV/FTC/TDF + Losartan | FTC/TDF + MK-0518 | FTC/TDF+MK-0518+Losartan
Number analyzed (Participants) | 12 | 10 | 10 | 10
participants | 12 | 10 | 10 | 10
Statistical Analysis 1: Comparison: EFV/FTC/TDF vs EFV/FTC/TDF + Losartan vs FTC/TDF + MK-0518 vs FTC/TDF+MK-0518+Losartan; Test type: Superiority; p = 1, Chi-squared, Corrected

9. Secondary Outcome: Changes in the CD4/CD8 Ratio in Peripheral Blood in Different Groups.
Time Frame: 48 weeks
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | EFV/FTC/TDF | EFV/FTC/TDF + Losartan | FTC/TDF + MK-0518 | FTC/TDF+MK-0518+Losartan
Number analyzed (Participants) | 12 | 10 | 10 | 10
ratio | -0.03 [-0.2 to 0.3] | 0.04 [-0.2 to 0.3] | 0.36 [0.0 to 0.5] | 0.37 [0.2 to 0.6]
Statistical Analysis 1: Comparison: EFV/FTC/TDF vs EFV/FTC/TDF + Losartan vs FTC/TDF + MK-0518 vs FTC/TDF+MK-0518+Losartan; Test type: Superiority; p = 0.01, Kruskal-Wallis

10. Secondary Outcome: Proportion of Patients With Reduced Intima-media Complex in Carotid Ultrasound in Different Groups.
Time Frame: 48 weeks
Population: Carotid ultrasound was performed at baseline in 41 out the 42 patients. However, only 36 patients repeated the ultrasound at week 48, and were included in the analysis (9 in each randomised group).
Measure: Number; unit: participants
Arm/Group | EFV/FTC/TDF | EFV/FTC/TDF + Losartan | FTC/TDF + MK-0518 | FTC/TDF+MK-0518+Losartan
Number analyzed (Participants) | 9 | 9 | 9 | 9
participants | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: EFV/FTC/TDF vs EFV/FTC/TDF + Losartan vs FTC/TDF + MK-0518 vs FTC/TDF+MK-0518+Losartan; Test type: Superiority; p = 1, Chi-squared, Corrected

11. Secondary Outcome: Proportion of Patients With Changes in Levels of Metalloproteinases
Time Frame: 48 weeks
Measure: Number; unit: participants
Arm/Group | EFV/FTC/TDF | EFV/FTC/TDF + Losartan | FTC/TDF + MK-0518 | FTC/TDF+MK-0518+Losartan
Number analyzed (Participants) | 12 | 10 | 10 | 10
participants | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: EFV/FTC/TDF vs EFV/FTC/TDF + Losartan vs FTC/TDF + MK-0518 vs FTC/TDF+MK-0518+Losartan; Test type: Superiority; p = 1, Chi-squared, Corrected

12. Secondary Outcome: Proportion of Patients With Changes in Levels of beta2-microglobulin.
Time Frame: 48 weeks
Measure: Number; unit: participants
Arm/Group | EFV/FTC/TDF | EFV/FTC/TDF + Losartan | FTC/TDF + MK-0518 | FTC/TDF+MK-0518+Losartan
Number analyzed (Participants) | 12 | 10 | 10 | 10
participants | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: EFV/FTC/TDF vs EFV/FTC/TDF + Losartan vs FTC/TDF + MK-0518 vs FTC/TDF+MK-0518+Losartan; Test type: Superiority; p = 1, Chi-squared, Corrected

13. Secondary Outcome: Proportion of Patients With Changes in Levels of CSF Cells.
Time Frame: 48 weeks
Measure: Number; unit: participants
Arm/Group | EFV/FTC/TDF | EFV/FTC/TDF + Losartan | FTC/TDF + MK-0518 | FTC/TDF+MK-0518+Losartan
Number analyzed (Participants) | 12 | 10 | 10 | 10
participants | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: EFV/FTC/TDF vs EFV/FTC/TDF + Losartan vs FTC/TDF + MK-0518 vs FTC/TDF+MK-0518+Losartan; Test type: Superiority; p = 1, Chi-squared, Corrected

14. Secondary Outcome: Proportion of Patients With Changes in Levels of Proteins.
Time Frame: 48 weeks
Measure: Number; unit: participants
Arm/Group | EFV/FTC/TDF | EFV/FTC/TDF + Losartan | FTC/TDF + MK-0518 | FTC/TDF+MK-0518+Losartan
Number analyzed (Participants) | 12 | 10 | 10 | 10
participants | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: EFV/FTC/TDF vs EFV/FTC/TDF + Losartan vs FTC/TDF + MK-0518 vs FTC/TDF+MK-0518+Losartan; Test type: Superiority; p = 1, Chi-squared, Corrected

15. Secondary Outcome: Proportion of Patients With Improvement in Neuropsychological Test
Time Frame: 48 weeks
Measure: Number; unit: participants
Arm/Group | EFV/FTC/TDF | EFV/FTC/TDF + Losartan | FTC/TDF + MK-0518 | FTC/TDF+MK-0518+Losartan
Number analyzed (Participants) | 12 | 10 | 10 | 10
participants | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: EFV/FTC/TDF vs EFV/FTC/TDF + Losartan vs FTC/TDF + MK-0518 vs FTC/TDF+MK-0518+Losartan; Test type: Superiority; p = 1, Chi-squared, Corrected

16. Secondary Outcome: Number of Participants With Adverse Events and Laboratory Abnormalities in the Different Groups.
Time Frame: up to 48 weeks
Measure: Number; unit: participants
Arm/Group | EFV/FTC/TDF | EFV/FTC/TDF + Losartan | FTC/TDF + MK-0518 | FTC/TDF+MK-0518+Losartan
Number analyzed (Participants) | 12 | 10 | 10 | 10
participants | 6 | 6 | 3 | 6
Statistical Analysis 1: Comparison: EFV/FTC/TDF vs EFV/FTC/TDF + Losartan vs FTC/TDF + MK-0518 vs FTC/TDF+MK-0518+Losartan; Test type: Superiority; p = 0.49, Chi-squared, Corrected

17. Secondary Outcome: Changes in CD4 CD38+ HLADR+ (%)
Description: Marker of activation in CD4 T cells. This Outcome Measure is reporting a change in the percentage of CD4 CD38+ HLADR+ T cells at 48 months minus the percentage at 0 weeks (baseline)
Time Frame: 0, 48 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of CD4 T cells
Arm/Group | EFV/FTC/TDF | EFV/FTC/TDF + Losartan | FTC/TDF + MK-0518 | FTC/TDF+MK-0518+Losartan
Number analyzed (Participants) | 12 | 10 | 10 | 10
percentage of CD4 T cells | 2.3 [1.4 to 5.5] | 4 [2.6 to 4.4] | 1.8 [1 to 2.5] | 2.2 [1.6 to 3]
Statistical Analysis 1: Comparison: EFV/FTC/TDF vs EFV/FTC/TDF + Losartan vs FTC/TDF + MK-0518 vs FTC/TDF+MK-0518+Losartan; Test type: Superiority; p = 0.02, Kruskal-Wallis

ADVERSE EVENTS:
Arm/Group | EFV/FTC/TDF | EFV/FTC/TDF + Losartan | FTC/TDF + MK-0518 | FTC/TDF+MK-0518+Losartan
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 6/12 | 6/10 | 3/10 | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EFV/FTC/TDF (N=12) | EFV/FTC/TDF + Losartan (N=10) | FTC/TDF + MK-0518 (N=10) | FTC/TDF+MK-0518+Losartan (N=10)
Post lumbar puncture headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) — Post lumbar puncture headache
Hepatitis C (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
High Blood Pressure (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendinitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver tests abonormalities (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sexual transmitted diseases (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Asthenia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gynecomastia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysthimia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes